CLINICAL TRIAL: NCT04527965
Title: Liver Fat as a Dietary Target for Treating Cardiometabolic Disorders in Prediabetes and Type 2 Diabetes: a Randomized Study (NAFLDiet)
Brief Title: Liver Fat as a Dietary Target for Treating Cardiometabolic Disorders in Prediabetes and Type 2 Diabetes
Acronym: NAFLDiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAFLDiet
Record Dates: First submitted 2020-08-05; First posted 2020-08-27 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: NAFLD; Diabetes Mellitus, Type 2; PreDiabetes
Keywords: NAFLD; Diabetes Mellitus, Type 2; Prediabetes; Fatty acids; Diet; Lipogenesis; Cardiometabolic risk
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Customized diet to reduce liver fat (Experimental): Ad libitum diet high in plant-derived PUFA and lower in carbohydrates
  Interventions: Other: Customized diet to reduce liver fat
- Healthy Nordic diet (Experimental): Ad libitum diet, based on Nordic foods, higher in carbohydrates (high fiber/low GI) and lower in fat but rich in monounsaturated fatty acids (MUFA) and PUFA
  Interventions: Other: Healthy Nordic diet
- Control (Active Comparator): Ad libitum diet in accordance with the Nordic Nutrition Recommendations
  Interventions: Other: Control

INTERVENTIONS:
Other: Customized diet to reduce liver fat — Ad libitum diet high in plant-derived PUFA and lower in carbohydrates
  Carbohydrates: 30 E% Fat: 50 E% (PUFA 10-15 E%) Protein: 20 E%
  Key foods are provided
  Arms: Customized diet to reduce liver fat
Other: Healthy Nordic diet — Ad libitum diet, based on Nordic foods, high in carbohydrates (high fiber/low GI) and lower in fat
  Carbohydrates: 50-55 E% Fat: 25-30 E% (PUFA 5-7.5 E%) Protein: 20 E%
  Key foods are provided
  Arms: Healthy Nordic diet
Other: Control — Ad libitum diet in accordance with the Nordic Nutrition Recommendations
  Key foods are provided
  Arms: Control

SUMMARY:
The overall aim of this study is to investigate the long-term impact of a customized diet aimed at reducing liver fat specifically and a healthy Nordic diet on ectopic fat (liver, pancreatic and visceral) and cardiometabolic risk in individuals with prediabetes and type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Randomized controlled studies investigating the impact of replacing dietary carbohydrates with polyunsaturated fat (PUFA) on liver fat content and cardiometabolic risk in individuals with prediabetes and T2D are lacking. Also, the effects of a Healthy Nordic Diet on liver fat content and glycemic control have not be investigated. This study therefore aims to:

* Investigate the effects of the diets on liver fat content (primary aim)
* Investigate the effects of the diets on pancreatic fat, visceral fat, lean tissue, glycemic and lipid control
* Investigate the effects of the diets on plasma markers of de novo lipogenesis (DNL) and desaturation (i.e. stearoyl-Coenzyme desaturase 1, SCD-1) as well as on hepatic DNL using MRI spectroscopy
* Investigate gene-diet interactions, especially if common gene variants (e.g. in PNPLA3) known to increase liver fat and dyslipidemia, may modify the dietary effects.
* Perform lipidomic analyses to identify potential mechanistic pathways that may associate with diet-induced changes in liver fat, pancreatic fat, visceral fat, insulin sensitivity, dyslipidemia or DNL

Our hypothesis is that a customized diet will effectively reduce liver fat through suppression of hepatic DNL and SCD-1 activity, and thereby improve atherogenic dyslipidemia, insulin resistance and hyperglycemia in individuals with prediabetes and T2D.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 30-75 years
* BMI 25-40
* T2D (duration ≤10 years, no insulin treatment) or prediabetes (ADA definition 2019) without diagnosed cardiovascular disease (CVD) during the last 2 years (e.g. myocardial infarction, stroke or angina pectoris)

Exclusion Criteria:

* BMI >40
* Alcohol intake >20 g/day
* Unwillingness to follow a new prescribed diet for 1 year
* Diet-induced weight loss (≥10%) the preceding 3 months of screening
* Malignant disease
* Severe kidney and liver disease
* Heart failure or other severe CVD
* claustrophobia or metal parts in the body (MRI)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Between-group changes in liver fat content between baseline and month 12 | 12 months
  Assessed by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Between-group changes in visceral adipose tissue mass between baseline and month 12 | 12 months
  Assessed by magnetic resonance imaging (MRI)
Between-group changes in lean tissue mass between baseline and month 12 | 12 months
  Assessed by magnetic resonance imaging (MRI)
Between-group changes in total body fat mass between baseline and month 12 | 12 months
  Assessed by magnetic resonance imaging (MRI)
Between-group changes in body weight between baseline and month 12 | 12 months
  Assessed by using a Tanita bioelectrical impedance analysis (BIA) scale
Between-group changes in glycated hemoglobin (HbA1c) between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry
Between-group changes in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry
Between-group changes in fasting plasma glucose between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry
Between-group changes in fasting serum insulin between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry
Between-group changes in systolic blood pressure between baseline and month 12 | 12 months
  Assessed by using an automated blood pressure monitor
Between-group changes in diastolic blood pressure between baseline and month 12 | 12 months
  Assessed by using an automated blood pressure monitor
Between-group changes in plasma lipids (total cholesterol, LDL cholesterol, triglycerides, HDL cholesterol, apoB and apoA1) between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry
Between-group changes in circulating inflammatory markers (CRP, Tumor Necrosis Factor Alpha-receptor 1 and 2, Interleukin-1 receptor antagonist, Fibroblast growth factor 21) between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry and ELISA
Between-group changes in pancreatic fat between baseline and month 12 | 12 months
  Assessed by magnetic resonance imaging (MRI)
Between-group changes in flow-mediated dilation (FMD) between baseline and month 12 | 12 months
  Assessed by ultrasound in approximately half of the study population (n=75)
Between-group changes in pulse-wave velocity (PWV) between baseline and month 12 | 12 months
  Assessed by ultrasound in approximately half of the study population (n=75)
Between-group values in FMD at month 12 | 12 months
  Assessed by ultrasound in the whole population (n=150)
Between-group values in PWV at month 12 | 12 months
  Assessed by ultrasound in the whole population (n=150)
Between-group changes in liver fat in prespecified subgroups and in individuals with low respectively high dietary compliance based on dietary and lipogenic biomarkers changes between baseline and month 12 | 12 months
  Assessed by magnetic resonance imaging (MRI)
Between-group changes in HbA1c in prespecified subgroups and in individuals with low respectively high dietary compliance based on dietary and lipogenic biomarkers changes between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry
Between-group changes in blood lipids in prespecified subgroups and in individuals with low respectively high dietary compliance based on dietary and lipogenic biomarkers changes between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry
Between-group changes in FIB-4 between baseline and month 12 | 12 months
  Assessed by routine clinical chemistry in combination with age

OTHER OUTCOMES:
Between-group changes in plasma-derived fatty acids and fatty acid ratios in the lipogenic pathway between baseline and month 12 | 12 months
  Assessed by gas chromatography (GC)
Between-group changes in imaging-derived fatty acids and fatty acid ratios in the lipogenic pathway between baseline and month 12 | 12 months
  Assessed by proton magnetic resonance spectroscopy (1 H-MRS)
Between-group changes in plasma lipids (ceramides) using a targeted lipidomic approach between baseline and month 12 | 12 months
  Lipids are measured using ultra-high performance liquid chromatography coupled to tandem mass spectrometry (UPLC-MS/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Risérus, PhD, Principal Investigator — Uppsala University; Lars Lind, MD, Study Director — Uppsala University
Locations (1):
- Uppsala univeristy hospital, Uppsala, Sweden

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT04527965/SAP_000.pdf